CLINICAL TRIAL: NCT06393751
Title: A Randomized Phase 1/2 Trial Evaluating the Addition of Tolinapant to Weekly Paclitaxel With or Without Bevacizumab in Patients With Recurrent Epithelial Ovarian Cancer
Brief Title: Testing the Addition of ASTX660 (Tolinapant) to the Usual Chemotherapy Treatment (Paclitaxel With or Without Bevacizumab) in Patients With Recurrent Ovarian Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Other - Protocol moved to Withdrawn
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-03344; NCI-2024-03344 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GY034 (Other: NRG Oncology); NRG-GY034 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2024-04-30; First posted 2024-05-01 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Platinum-Refractory Fallopian Tube Carcinoma; Platinum-Refractory Ovarian Carcinoma; Platinum-Refractory Primary Peritoneal Carcinoma; Recurrent Fallopian Tube Adenocarcinoma; Recurrent Fallopian Tube Carcinosarcoma; Recurrent Fallopian Tube Clear Cell Adenocarcinoma; Recurrent Fallopian Tube High Grade Serous Adenocarcinoma; Recurrent Fallopian Tube Undifferentiated Carcinoma; Recurrent High Grade Endometrioid Adenocarcinoma; Recurrent Ovarian Adenocarcinoma; Recurrent Ovarian Carcinosarcoma; Recurrent Ovarian Clear Cell Adenocarcinoma; Recurrent Ovarian High Grade Serous Adenocarcinoma; Recurrent Ovarian Seromucinous Carcinoma; Recurrent Ovarian Undifferentiated Carcinoma; Recurrent Platinum-Resistant Fallopian Tube Carcinoma; Recurrent Platinum-Resistant Ovarian Carcinoma; Recurrent Platinum-Resistant Primary Peritoneal Carcinoma; Recurrent Primary Peritoneal Adenocarcinoma; Recurrent Primary Peritoneal Carcinosarcoma; Recurrent Primary Peritoneal Clear Cell Adenocarcinoma; Recurrent Primary Peritoneal High Grade Serous Adenocarcinoma; Recurrent Primary Peritoneal Undifferentiated Carcinoma
MeSH Terms: interventions — Bevacizumab; Immunoglobulin G; Disulfides; Specimen Handling; Magnetic Resonance Spectroscopy; Paclitaxel; Taxes; ASTX-660

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase I (paclitaxel, tolinapant, bevacizumab) (Experimental): Patients receive paclitaxel IV on days 1, 8 and 15, bevacizumab IV on days 1 and 15, and ASTX660 PO on days 1-7 and 15-21 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection, CT and MRI throughout the study.
  Interventions: Biological: Bevacizumab; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Paclitaxel; Drug: Tolinapant
- Phase II, Arm I (paclitaxel, bevacizumab) (Active Comparator): Patients receive paclitaxel IV on days 1, 8, and 15 of each cycle. Patients may also receive bevacizumab IV on days 1 and 15 of each cycle per provider. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection, CT and MRI throughout the study.
  Interventions: Biological: Bevacizumab; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Paclitaxel
- Phase II, Arm II (paclitaxel, tolinapant, bevacizumab) (Experimental): Patients receive paclitaxel IV on days 1, 8, and 15 and ASTX660 PO on days 1-7 and 15-21 of each cycle. Patients may also receive bevacizumab IV on days 1 and 15 of each cycle per provider. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection, CT and MRI throughout the study.
  Interventions: Biological: Bevacizumab; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Paclitaxel; Drug: Tolinapant

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Drug: Tolinapant — Given PO
  Other Names: ASTX 660; ASTX660; XIAP/cIAP1 Antagonist ASTX660
  Arms: Phase I (paclitaxel, tolinapant, bevacizumab); Phase II, Arm II (paclitaxel, tolinapant, bevacizumab)

SUMMARY:
This phase I/II trial tests the safety, best dose and effectiveness of adding tolinapant (ASTX660) to paclitaxel with or without bevacizumab in treating patients with ovarian cancer that has come back after a period of improvement (recurrent). Tolinapant may stop the growth of tumor cells by blocking proteins, such as XIAP and cIAP1, that promote the growth of tumor cells and increase resistance to chemotherapy. Paclitaxel is in a class of medications called antimicrotubule agents. It stops tumor cells from growing and dividing and may kill them. Bevacizumab is in a class of medications called antiangiogenic agents. It works by stopping the formation of blood vessels that bring oxygen and nutrients to the tumor. This may slow the growth and spread of tumor cells. Adding ASTX660 to paclitaxel with or without bevacizumab may be safe, tolerable and/or effective in treating patients with recurrent ovarian cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of adding ASTX660 (tolinapant) to a regimen of weekly paclitaxel with bevacizumab. (Phase I) II. To determine the recommended phase 2 dose (RP2D) for the combination of ASTX660 (tolinapant) and weekly paclitaxel with bevacizumab. (Phase I) III. To assess the efficacy of adding ASTX660 (tolinapant) to weekly paclitaxel, with or without bevacizumab (investigator choice), as measured by progression free survival (PFS). (Phase II)

SECONDARY OBJECTIVES:

I. To assess the objective response rate (ORR) of the addition of ASTX660 (tolinapant) to weekly paclitaxel with or without bevacizumab as compared to weekly paclitaxel with or without bevacizumab.

II. To assess overall survival.

EXPLORATORY OBJECTIVE:

I. To explore whether lack of cIAP1 expression results in no benefit for the addition of ASTX660 (tolinapant) to weekly paclitaxel +/- bevacizumab.

OUTLINE: This is a phase I, dose escalation study of ASTX660 and paclitaxel with or without bevacizumab followed by a dose expansion study. The phase II study will follow completion of the phase I study.

PHASE I:

Patients receive paclitaxel intravenously (IV) on days 1, 8 and 15, bevacizumab IV on days 1 and 15, and ASTX660 orally (PO) on days 1-7 and 15-21 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection, computed tomography (CT) and magnetic resonance imaging (MRI) throughout the study.

PHASE II: Patients are randomized to 1 of 2 arms.

ARM I (CONTROL): Patients receive paclitaxel IV on days 1, 8, and 15 of each cycle. Patients may also receive bevacizumab IV on days 1 and 15 of each cycle per provider. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection, CT and MRI throughout the study.

ARM II (EXPERIMENTAL): Patients receive paclitaxel IV on days 1, 8, and 15 and ASTX660 PO on days 1-7 and 15-21 of each cycle. Patients may also receive bevacizumab IV on days 1 and 15 of each cycle per provider. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection, CT and MRI throughout the study.

After completion of study treatment, patients are followed up every 3 months for 2 years then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of high grade epithelial ovarian, fallopian tube, or primary peritoneal cancer. Required: submission of pathology report

  * Patients with the following histologic cell types are eligible:

    * High grade serous
    * Endometrioid, grade 3
    * Clear cell
    * Undifferentiated
    * Mixed epithelial
    * Carcinosarcoma
    * Adenocarcinoma, not otherwise specified (NOS)
* Patients must be considered to have platinum-resistant or platinum-refractory recurrent ovarian cancer to be enrolled in this trial

  * Platinum-resistant disease is defined as progression within < 6 months from completion of platinum-based therapy. The date should be calculated from the last administered dose of platinum therapy
  * Platinum-refractory disease is defined as progression within 30 days of completing the last dose of platinum during initial therapy. The date should be calculated from the last administered dose of platinum therapy
* Patients must have evaluable disease or measurable disease defined by Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded). Each lesion must be ≥ 10 mm when measured by CT or MRI. Lymph nodes must be ≥ 15 mm in short axis when measured by CT or MRI. Previously irradiated lesions can be considered as measurable disease only if progressive disease has been unequivocally documented at that site since radiation
* Patients with treated brain metastases are eligible if follow up brain imaging after central nervous system (CNS) directed therapy shows no evidence of progression
* Patients must have received ≥ 1 platinum-based therapy and not more than 5 prior lines of therapies. Notes:

  * Adjuvant/neoadjuvant therapy is counted as only 1 regimen in the absence of intervening progression.
  * Maintenance therapy (e.g., bevacizumab, poly adenosine diphosphate-ribose polymerase [PARP] inhibitor will be considered part of the preceding line of therapy [i.e., not counted independently])
  * Therapy changed due to toxicity in the absence of progression will be considered part of the same line (i.e., not counted independently)
  * Hormonal therapy will not be counted as a separate line of therapy
* Age ≥ 18
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Absolute neutrophil count (ANC) ≥ 1,500 cells/mm^3
* Platelets ≥ 100,000 cells/mm^3
* Hemoglobin ≥ 8 g/dl
* Creatinine ≤ institutional upper limit of normal (ULN), OR calculated creatinine clearance (CrCL) of ≥ 50 mL/min by the Cockcroft-Gault formula
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (patients with known Gilbert's disease who have bilirubin level ≤ 3 x ULN may be enrolled)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x institutional ULN
* Patients with a known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry and, for patients treated in the United States (U.S.), authorization permitting release of personal health information
* No active infection requiring parental antibiotics
* No evidence of intra-abdominal abscess, abdominal/pelvic fistula, gastrointestinal perforation, gastrointestinal (GI) obstruction, and/or with drainage gastrostomy tube required. NOTE: required interval since last bowel obstruction: 30 day minimum for incomplete obstruction, resolved with conservative means; 6 months for fistula

Exclusion Criteria:

* Patients who have received prior weekly paclitaxel in a platinum-resistant setting
* Major surgical procedure within 28 days prior to registration, or anticipation of need for major surgical procedure during the study. Note: Placement of a vascular access device, thoracentesis, and/or paracentesis will not be considered major surgery
* Women who are pregnant or are unwilling to discontinue nursing
* Evidence of bleeding diathesis or clinically significant coagulopathy within the past 3 months. Patients are not excluded for past or current use of anticoagulation
* Uncontrolled hypertension (systolic blood pressure [SBP] > 150 and/or diastolic blood pressure [DBP] > 90)
* Patients currently taking and unwilling/unable to discontinue the use of drugs that are known to inhibit or induce P-glycoprotein (gp)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-10-31 (Estimated); Primary Completion 2028-02-09 (Estimated); Study Completion 2028-02-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (Phase I) | At 28 days
  Assessed using the Bayesian Optimal Interval design. Toxicity will be graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0.
Progression free survival (PFS) (Phase II) | At randomization to progressive disease or death, assessed up to 5 years after completion of study treatment
  The primary hypothesis test will be based on a logrank test, stratified on factors declared at randomization. The PFS hazard ratio will be estimated by Cox regression, stratified by factors declared at randomization. The treatment hazard ratio estimates and their 95% confidence intervals will be estimated using proportional hazards models specified to be consistent with the logrank tests.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 30 days after last dose of study treatment
  AEs will be defined as any untoward medical occurrence associated wtih the use of a drug in humans, whether or not considered drug related. AEs will be graded using NCI CTCAE v5.0. All AEs will be summarized.
Overall survival (OS) | At randomization to death, assessed up to 5 years after completion of study treatment
  OS will be defined as the time from randomization to death from any cause. The OS treatment hypothesis will be based on a logrank test, stratified by the factors specified at randomization. Comparisons of the OS distributions by treatment arm will be described using Kaplan-Meier methods. Treatment hazard ratio estimates and their 95% confidence intervals will be estimated using a multivariable proportional hazards model specified with main effects for the randomization treatment assignment and stratified by the factors declared at randomization.
Objective response rate (ORR) | At start of treatment to disease progression/recurrence, assessed up to 5 years after completion of treatment
  ORR will be defined as the binomial proportion of evaluable patients with a best overall response of complete response (CR) or partial response (PR) by Response Evaluation Criteria in Solid Tumors. The ORR estimates by treatment arm will be supported by their 2-sided, 95% Wilson-Score confidence intervals. The relative odds of response in the experimental arm will be estimated using a multivariable logistic regression model specified with main effects for the treatment groups and stratified by the stratification factors reported at baseline.
Duration of response (DOR) | At first response to progression or death, assessed up to 5 years after completion of study treatment
  DOR will be defined as the time from first documentation of either PR or CR until disease progression or death, whichever is observed first. Treatment group differences in response duration will be graphed using Kaplan-Meier methods and compared using logrank tests, stratified by the factors declared at randomization. The relative hazards of progression or death in each group will be estimated using similarly stratified proportional hazards regression model specified with main effects for the treatment indicator.

OTHER OUTCOMES:
Lack of cIAP1 expression | Up to 5 years after completion of study treatment
  Will evaluate whether lack of cIAP1 expression results in no benefit for the addition of ASTX660 to weekly paclitaxel. The null hypothesis of no predictive effect of cIAP1 on clinical outcomes will be assessed using the type 3 score test for the interaction of the randomized treatment assignment and the patient-level cIAP1 histopathological-score classification (positive, reference negative). The type 3 test result will be obtained from a multivariable Cox regression model model specified with main effects for the randomized treatment assignment and the cIAP1 classification (negative/positive), and the interaction term. The model may be stratified by bevacizumab use. Treatment hazard ratios and 95% confidence intervals will be estimated within the cIAP1 subgroups, and graphed in a forest plot to assess qualitative interactions.
ORR (Phase I/Ib) | Up to 5 years after completion of study treatment
  ORR will be compared among patients enrolled in the phase I/Ib parts of the trial. Treatment effect estimates of clinical benefit will be descriptive.
PFS (Phase I/Ib) | Up to 6 months after starting treatment
  PFS will be compared among patients enrolled in the phase I/Ib parts of the trial. Treatment effect estimates of clinical benefit will be descriptive. Dose level effects on PFS will be described using Kaplan Meier methods. Treatment effectiveness will be quantified using estimates for the proportion of patients who are alive without documented progression 6 months after starting treatment.
OS (Phase I/Ib) | Up to 6 months after starting treatment
  OS will be compared among patients enrolled in the phase I/Ib parts of the trial. Treatment effect estimates of clinical benefit will be descriptive. Dose level effects on oS will be described using Kaplan Meier methods. Treatment effectiveness will be quantified using estimates for the proportion of patients who are alive 6 months after starting treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen P Zeligs, Principal Investigator — NRG Oncology

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm